CLINICAL TRIAL: NCT06761066
Title: 36-week, Single-center, Randomized, Double-blind, Parallel-design, Placebo-controlled Trial to Determine the Safety and Efficacy of NVP-NK4146 in Patients with Mild Cognitive Impairment (MCI) Due to Alzheimer's Disease
Brief Title: Efficacy and Safety of NVP-NK4146 in Patients with Mild Cognitive Impairment (MCI) Due to Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NVP-NK4146_HS
Record Dates: First submitted 2024-12-17; First posted 2025-01-07 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Group (Experimental): NVP-NK4146
  Interventions: Dietary Supplement: NVP-NK4146
- Placebo Group (Placebo Comparator): NVP-NK4146 Placebo
  Interventions: Dietary Supplement: NVP-NK4146 Placebo

INTERVENTIONS:
Dietary Supplement: NVP-NK4146 — BID for 36 weeks orally
  Arms: Active Group
Dietary Supplement: NVP-NK4146 Placebo — BID for 36 weeks orally
  Arms: Placebo Group

SUMMARY:
The purpose of this clinical trial is to exploratively evaluate the efficacy and safety of NVP -NK4146 in improving mild cognitive impairment (MCI) in patients with due to Alzheimer's disease (AD) compared to placebo

DETAILED DESCRIPTION:
36-week, single-center, randomized, double-blind, parallel-design, placebo-controlled trial

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 60 or older
2. Subject who meet the National Institute of Aging and Alzheimer's Associations (NIA-AA) core clinical criteria for MCI and have positive readings from amyloid PET
3. Subject who can read and understand the Informed Consent Form and legends and who voluntarily decided to participate in current clinical trial and have signed the Informed Consent Form

Exclusion Criteria:

1. Subject diagnosed with dementia according to the criteria of DSM-5 or ICD-10
2. Subject currently receiving treatment for malignant tumors (except those who have fully recovered from cancer for more than 5 years or those with basal cell carcinoma, squamous cell carcinoma, or prostate cancer may participate at the investigator's discretion)
3. Subject who are illiterate and/or without any education
4. Any other factors deemed by the investigator to be likely to ineligible for the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
amyloid PET scan | baseline and 36 weeks
  Changes in brain amyloid measured by amyloid PET scan from baseline to 36 weeks

SECONDARY OUTCOMES:
ADAS-Cog(Alzheimer's Disease Assessment Scale-Cognitive Subscale)13 | baseline and 36 weeks
  Changes in ADAS-Cog 13 total score, memory score, and subscales from baseline to 36 weeks
CDR-SB(Clinical Dementia Rating-Sum of Boxes) | baseline and 36 weeks
  Changes in CDR-SB(Clinical Dementia Rating-Sum of Boxes) and CDR total score from baseline to 36 weeks
GDS (Global Deterioration Scale) | baseline and 36 weeks
  Change in GDS total score from baseline to 36 weeks
K-MMSE (the Korean Mini-Mental State Examination) | baseline and 36 weeks
  Change in K-MMSE total score from baseline to 36 weeks

IPD SHARING:
Plan to Share IPD: No